CLINICAL TRIAL: NCT00970502
Title: Phase I/II Dose Escalation Trial of Induction and Concomitant Erlotinib and Celecoxib With Radiation Therapy for Treatment of Poor Prognosis Head and Neck Cancer, Including Reirradiation
Brief Title: Erlotinib, Celecoxib and Reirradiation for Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johnny Kao (Other)
Responsible Party: Sponsor-Investigator, Johnny Kao, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 06-0509
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Cancer of the Pharynx; Cancer of the Larynx; Cancer of the Neck; Paranasal Sinus Neoplasms; Cancer of the Head
Keywords: celecoxib; erlotinib; epidermal growth factor receptor; intensity-modulated radiotherapy; cyclooxygenase-2; reirradiation
MeSH Terms: conditions — Pharyngeal Neoplasms; Laryngeal Neoplasms; Head and Neck Neoplasms; Paranasal Sinus Neoplasms | interventions — Erlotinib Hydrochloride; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- erlotinib + celecoxib (Experimental)
  Interventions: Drug: erlotinib + celecoxib

INTERVENTIONS:
Drug: erlotinib + celecoxib — In this phase I/II study, patients will be treated with daily erlotinib 150 mg and twice-daily celecoxib 200 to 600 mg for 14 days. Re-irradiation with IMRT will start on day 15 and will continue for 5.5 to 6.5 weeks along with erlotinib and celecoxib. After completion of radiation, patients will be given the option of continuing on erlotinib for 2 years or until unacceptable toxicity or disease progression
  Other Names: Tarceva; Celebrex

SUMMARY:
There is no optimal treatment for patients with recurrent head and neck cancer after previous radiation. Chemotherapy alone is not curative and patients survive an average of only 6 to 10 months. Surgery is not always possible and often cannot remove every cancerous cell. On the other hand, reirradiation with chemotherapy cures approximately 25 to 30% of patients but has significant toxicity with as many as 15 to 20% suffering from life-threatening or fatal complications. Therefore, less toxic and more effective reirradiation regimens are urgently needed. There are extensive data from animal studies and preliminary human studies showing that blocking epidermal growth factor receptor (EGFR) and COX-2 enhances radiation effect and is more effective than either treatment alone. Erlotinib is a FDA approved oral inhibitor of EGFR and celecoxib is a FDA approved COX-2 inhibitor. Both have been well studied in humans and appear to have less severe toxicity than conventional chemotherapeutic agents.

DETAILED DESCRIPTION:
Despite advances in the treatment of head and neck cancer, locoregional recurrences are the predominant site of treatment failure and are frequently the cause of death. Second primary tumors in the head and neck occur in up to 30% of patients at 10 years of follow-up after eradication of the original tumor due to field cancerization. The standard approach to patients with recurrent but non-metastatic disease has been surgical salvage alone. Unfortunately, this strategy is feasible in only a select group of patients and 5 year survival rates have ranged from 15-40%.

Most patients with previously irradiated unresectable recurrent or metastatic head and neck cancer are treated with chemotherapy alone. This approach has offered limited palliation with response rates of 10-40%, median survival of 5 to 10 months. While this may be an acceptable option for patients with clearly incurable widespread metastatic disease, it may not be the best approach for those patients with potentially curable locoregional disease.

While geographic misses and second primary tumors occur, the majority of patients have radioresistant tumors. Therefore, reirradiation alone is unlikely to be effective. High dose reirradiation with concomitant chemotherapy represents a more aggressive approach resulted in encouraging 3-year survival rates of 15 to 35%. This approach represents a potentially curative option for patients with unresectable or partially resected disease arising in a previously irradiated volume. However, the high rates of acute and late toxicity with this approach have limited widespread application of this approach.

Extensive preclinical and clinical data suggest that both epidermal growth factor receptor (EGFR) antagonists and cyclooxygenase-2 (COX-2) inhibitors enhance the effectiveness of ionizing radiation. In locally advanced head and neck cancer, a recent phase III trial concurrent anti-EGFR monoclonal antibody and radiation demonstrated improved local control, disease free survival and overall survival compared to radiation alone without the increased mucosal toxicity associated with concurrent chemotherapy. COX-2 inhibition and anti-EGFR therapy demonstrates activity against recurrent/metastatic head and neck cancer in a recent phase I study. Head and neck cancer represents an ideal site to study biologic markers of tumor response because of the accessibility of tumors for biopsy. Therefore, we propose the combination of Erlotinib and Celecoxib with radiation in a cohort of previously irradiation patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologically or cytologically confirmed diagnosis of squamous cell or poorly differentiated carcinomas of the head and neck or lymphoepithelioma
* Prior radiation to the head and neck, surgery or chemotherapy is allowed
* Karnofsky performance status of >= 70%
* Intact organ and bone marrow function
* Obtained informed consent

Exclusion Criteria:

* Demonstration of metastatic disease (i.e. M1 disease).
* Incomplete healing from previous surgery
* Pregnancy or breast feeding (men and women of child-bearing potential are eligible but must consent to using effective contraception during therapy and for at least 3 months after completing therapy)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with clinically significant pulmonary dysfunction, cardiomyopathy, or any history of clinically significant CHF are excluded. The exclusion of patients with active coronary artery disease will be at the discretion of the attending physician.
* Uncontrolled active infection unless curable with treatment of their cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Kao, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Salama JK, Vokes EE, Chmura SJ, Milano MT, Kao J, Stenson KM, Witt ME, Haraf DJ. Long-term outcome of concurrent chemotherapy and reirradiation for recurrent and second primary head-and-neck squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2006 Feb 1;64(2):382-91. doi: 10.1016/j.ijrobp.2005.07.005. Epub 2005 Oct 5. PMID 16213104
- [Background] Kao J, Garofalo MC, Milano MT, Chmura SJ, Citron JR, Haraf DJ. Reirradiation of recurrent and second primary head and neck malignancies: a comprehensive review. Cancer Treat Rev. 2003 Feb;29(1):21-30. doi: 10.1016/s0305-7372(02)00096-8. PMID 12633577
- [Background] J. Kao, S. H. Packer, M. Teng, V. Gupta, K. Misiukiewicz, E. M. Genden; Mount Sinai School of Medicine, New York, NY, J Clin Oncol 28:15s, 2010 (suppl; abstr 5561).
- [Result] Kao J, Genden EM, Chen CT, Rivera M, Tong CC, Misiukiewicz K, Gupta V, Gurudutt V, Teng M, Packer SH. Phase 1 trial of concurrent erlotinib, celecoxib, and reirradiation for recurrent head and neck cancer. Cancer. 2011 Jul 15;117(14):3173-81. doi: 10.1002/cncr.25786. Epub 2011 Jan 18. PMID 21246519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were evaluated by head and neck surgery, medical oncology, and radiation oncology before trial entry. Patients were enrolled at least 6 months after they had completed prior radiation. Patients were enrolled between March 2007 and December 2009.
Period: Overall Study
Arm/Group | Erlotinib + Celecoxib
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 15 subjects consented, one withdrew before receiving study treatment and was excluded from analysis
Arm/Group | Erlotinib + Celecoxib
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 64 [43 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
ECOG Performance Status [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) 0 - Fully active, able to carry on all pre-disease performance without restriction
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature 2- Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  participants
    0 | 0
    1 | 5
    2 | 9
Tobacco use, pack-years [Number; unit: participants]
  None to minimal | 2
  <20 | 6
  20-40 | 3
  >40 | 2
  Unknown | 1
Recurrent vs secondary primary [Number; unit: participants]
  Primary recurrence | 7
  Second or later recurrence | 4
  Second primary cancer | 3
Histology [Number; unit: participants]
  Squamous cell carcinoma | 13
  Adenoid cystic | 1
Primary Site [Number; unit: participants]
  Sinonasal | 3
  Ear/facial skin | 2
  Oropharynx | 3
  Oral cavity | 1
  Hypopharynx | 4
  Larynx | 1
Primary tumor classification [Number; unit: participants] — T4 --> Tumor of any size with direct extension to chest wall or skin Tx - T3 --> any tumor not classified as T4
  participants
    Tx-T3 | 4
    T4 | 10
Lymph node status [Number; unit: participants] — N0 - tumor cells absent from regional lymph nodes N1 - regional lymph node metastasis present; (at some sites; tumor spread to closest or small number of regional lymph nodes)
  participants
    N0 | 3
    N1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Number of participants with acute and late toxicity
Time Frame: 30 DAYS
Population: Erlotinib and celecoxib were administered orally
Measure: Number; unit: participants
Groups:
- Celecoxib 200mg: Dose Level 1: Patients administered 150mg Erlotinib daily and 200mg Celecoxib twice daily
- Celecoxib 400mg: Dose Level 2: Patients administered 150mg Erlotinib daily and 400mg Celecoxib twice daily
- Celecoxib 600mg: Dose Level 3: Patients administered 150mg Erlotinib daily and 600mg Celecoxib twice daily
Arm/Group | Celecoxib 200mg | Celecoxib 400mg | Celecoxib 600mg
Number analyzed (Participants) | 3 | 8 | 3
participants | 0 | 1 | 2

2. Secondary Outcome: Clinical Response
Description: Response to Concurrent Erlotinib, Celecoxib, and Reirradiation according to Response Evaluation Criteria in Solid Tumors - Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 20 months
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib + Celecoxib
Number analyzed (Participants) | 14
Participants
  Complete Response(CR) | 6
  Pathologic partial response (pPR) | 1
  Progressive disease (PD) | 5
  No evidence of disease (NED) | 2

3. Secondary Outcome: Locoregional Progression
Description: Patients with locoregional and/or distant progression
Time Frame: 20 months
Measure: Number; unit: participants
Arm/Group | Erlotinib + Celecoxib
Number analyzed (Participants) | 14
participants
  free of disease | 4
  isolated locoregional progression | 4
  isolated distant progression | 2
  both locoregional and distant progression | 1
  no evidence of disease, died of comorbid illness | 3

4. Secondary Outcome: Locoregional Control, Progression-free Survival, Overall Survival and Late Toxicity
Description: At a median follow-up of 11 months, the 1 year locoregional control, progression-free survival, and overall survival rates.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Groups:
- Erlotinib + Celecoxib: Recommended dose of celecoxib was 400mg
Arm/Group | Erlotinib + Celecoxib
Number analyzed (Participants) | 15
percentage of participants
  locoregional control | 60
  progress-free survival | 37
  overall survival rates | 55
  long term toxicity | 0

ADVERSE EVENTS:
Arm/Group | Erlotinib + Celecoxib
Serious Adverse Events (participants affected / at risk) | 14/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib + Celecoxib (N=14)
pharyngocutaneous fistula (Gastrointestinal disorders) | 1 (1)
folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
nausea (General disorders) | 1 (1)
rectal bleeding (Gastrointestinal disorders) | 1 (1)
bone necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Pain (General disorders) | 3
Fatigue (General disorders) | 2
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1
Metabolic (Na, K, Ca) (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Celecoxib (N=14)
Mucositis (Gastrointestinal disorders) | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 12
Pain (General disorders) | 11
Xerostomia (General disorders) | 5
abnormal white blood cell count (Blood and lymphatic system disorders) | 5
abnormal hemoglobin count (Blood and lymphatic system disorders) | 12
Fatigue (General disorders) | 3
Dry eye (Eye disorders) | 1
Nausea (General disorders) | 1
Acneiform rash (Skin and subcutaneous tissue disorders) | 12
Metabolic (Na, K, Ca) (Metabolism and nutrition disorders) | 4
Elevated Liver Function Tests (Hepatobiliary disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
Conjuncitivitis (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes